CLINICAL TRIAL: NCT03960112
Title: Multicentric Evaluation of the True Negative Predictive Value of Multiparametric MRI for the Detection of Prostate Cancer Using Cystoprostatectomy Specimen as Reference
Acronym: NPV-MRI-02
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Institut Paoli-Calmettes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NPV-MRI-02-IPC 2017-047
Record Dates: First submitted 2018-09-18; First posted 2019-05-22 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Prostate Cancer
Keywords: multiparametric MRI; cystoprostatectomy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Multiparametric Magnetic Resonance Imaging

STUDY DESIGN:
Intervention Model Description: Per patient analysis in a prospective, multicenter cohort, open study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- mpMRI (Experimental): mpMRI in the detection of prostate cancer in a per patient analysis using cystoprostatectomy specimen
  Interventions: Device: mpMRI

INTERVENTIONS:
Device: mpMRI — mpMRI in the detection of prostate cancer in a per patient analysis using cystoprostatectomy specimen

SUMMARY:
To evaluate the negative predictive value of mpMRI in the detection of prostate cancer using cystoprostatectomy specimen as the reference

DETAILED DESCRIPTION:
To evaluate the negative predictive value of mpMRI in the detection of prostate cancer using cystoprostatectomy specimen as the reference

ELIGIBILITY:
Inclusion Criteria:

1. age >18 years
2. male patient scheduled for cystoprostatectomy as treatment of muscle invasive bladder cancer (clinical T2-T3, any N) or high risk non-muscle invasive bladder cancer (pT1 or CIS)
3. no known diagnosis of prostate cancer
4. no contraindication to undergo multiparametric MRI
5. Signed written informed consent prior to any screening procedures being performed
6. Patient affiliated to the ''National security'' regimen or beneficiary of this regimen

Exclusion Criteria:

1. allergy against MR contrast media
2. diagnosis or previous treatment of prostate cancer
3. severe renal insufficiency (GFR <30ml/min)
4. Bladder cancer infiltrating the prostate (T4)
5. Pelvic metallic implants such as hip prosthesis
6. Patients scheduled for cystoprostatectomy with prostate capsule sparing
7. Patients unable to provide informed consent
8. Patients having a prostate biopsy <6 month

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — male patient scheduled for cystoprostatectomy as treatment of muscle invasive bladder cancer
Enrollment: 150 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2022-10-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Negative predictive value of mpMRI in the detection of prostate cancer using cystoprostatectomy specimen as the reference | From the date of mpMRI exam (Day-1) to the date pathology report of Day 0 surgery is obtained (an average of 7 days)
  The true negative and false negative rates of mpMRI in the detection of prostate cancer in a per patient analysis using cystoprostatectomy specimen as a reference in patients with no previous diagnosis of prostate cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Jochen WALZ, MD, Principal Investigator — Institut Paoli-Calmettes
Locations (5):
- France (5):
  - Institut Paoli Calmettes, Marseille, Bouches Du Rhone
  - CHRU Hopital Edouard Herriot, Lyon
  - Hopital Nord, Marseille
  - Institut Mutualiste Montsouris, Paris
  - Chu Saint Etienne, Saint-Etienne

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moldovan PC, Van den Broeck T, Sylvester R, Marconi L, Bellmunt J, van den Bergh RCN, Bolla M, Briers E, Cumberbatch MG, Fossati N, Gross T, Henry AM, Joniau S, van der Kwast TH, Matveev VB, van der Poel HG, De Santis M, Schoots IG, Wiegel T, Yuan CY, Cornford P, Mottet N, Lam TB, Rouviere O. What Is the Negative Predictive Value of Multiparametric Magnetic Resonance Imaging in Excluding Prostate Cancer at Biopsy? A Systematic Review and Meta-analysis from the European Association of Urology Prostate Cancer Guidelines Panel. Eur Urol. 2017 Aug;72(2):250-266. doi: 10.1016/j.eururo.2017.02.026. Epub 2017 Mar 21. PMID 28336078
- [Background] N. Mottet JB, E. Briers, R.C.N. van den Bergh, M. Bolla, N.J. van Casteren, P. Cornford, S. Culine, S. Joniau, T. Lam, M.D. Mason, V. Matveev, H. van der Poel, T.H. van der Kwast, O. Rouvière, T. Wiegel. Guidelines on prostate cancer. European Association of Urology Web site https://uroweborg/guideline/prostate-cancer/. Accessed May 17, 2016.
- [Background] Schoots IG, Petrides N, Giganti F, Bokhorst LP, Rannikko A, Klotz L, Villers A, Hugosson J, Moore CM. Magnetic resonance imaging in active surveillance of prostate cancer: a systematic review. Eur Urol. 2015 Apr;67(4):627-36. doi: 10.1016/j.eururo.2014.10.050. Epub 2014 Nov 15. PMID 25511988
- [Background] Le JD, Tan N, Shkolyar E, Lu DY, Kwan L, Marks LS, Huang J, Margolis DJ, Raman SS, Reiter RE. Multifocality and prostate cancer detection by multiparametric magnetic resonance imaging: correlation with whole-mount histopathology. Eur Urol. 2015 Mar;67(3):569-76. doi: 10.1016/j.eururo.2014.08.079. Epub 2014 Sep 23. PMID 25257029
- [Background] Branger N, Maubon T, Traumann M, Thomassin-Piana J, Brandone N, Taix S, Touzlian J, Brunelle S, Pignot G, Salem N, Gravis G, Walz J. Is negative multiparametric magnetic resonance imaging really able to exclude significant prostate cancer? The real-life experience. BJU Int. 2017 Mar;119(3):449-455. doi: 10.1111/bju.13657. Epub 2016 Oct 4. PMID 27618134
- [Background] Ahmed HU, El-Shater Bosaily A, Brown LC, Gabe R, Kaplan R, Parmar MK, Collaco-Moraes Y, Ward K, Hindley RG, Freeman A, Kirkham AP, Oldroyd R, Parker C, Emberton M; PROMIS study group. Diagnostic accuracy of multi-parametric MRI and TRUS biopsy in prostate cancer (PROMIS): a paired validating confirmatory study. Lancet. 2017 Feb 25;389(10071):815-822. doi: 10.1016/S0140-6736(16)32401-1. Epub 2017 Jan 20. PMID 28110982
- [Background] Robertson NL, Hu Y, Ahmed HU, Freeman A, Barratt D, Emberton M. Prostate cancer risk inflation as a consequence of image-targeted biopsy of the prostate: a computer simulation study. Eur Urol. 2014 Mar;65(3):628-34. doi: 10.1016/j.eururo.2012.12.057. Epub 2013 Jan 3. PMID 23312572
- [Background] Wetterauer C, Weibel M, Gsponer JR, Vlajnic T, Zellweger T, Butikofer S, Muller G, Puschel H, Bachmann A, Gasser TC, Bubendorf L, Rentsch CA. Incidental prostate cancer prevalence at radical cystoprostatectomy--importance of the histopathological work-up. Virchows Arch. 2014 Dec;465(6):629-36. doi: 10.1007/s00428-014-1656-9. Epub 2014 Oct 1. PMID 25269630
- [Background] Bains LJ, Studer UE, Froehlich JM, Giannarini G, Triantafyllou M, Fleischmann A, Thoeny HC. Diffusion-weighted magnetic resonance imaging detects significant prostate cancer with high probability. J Urol. 2014 Sep;192(3):737-42. doi: 10.1016/j.juro.2014.03.039. Epub 2014 Mar 15. PMID 24641913
- [Background] Steinberg DM, Fine J, Chappell R. Sample size for positive and negative predictive value in diagnostic research using case-control designs. Biostatistics. 2009 Jan;10(1):94-105. doi: 10.1093/biostatistics/kxn018. Epub 2008 Jun 12. PMID 18556677
- [Background] DeLong ER, DeLong DM, Clarke-Pearson DL. Comparing the areas under two or more correlated receiver operating characteristic curves: a nonparametric approach. Biometrics. 1988 Sep;44(3):837-45. PMID 3203132